CLINICAL TRIAL: NCT06663748
Title: Evaluate the Efficacy and Safety of ARX788 Given Every 6 Weeks in Patients with HER2-positive Advanced Breast Cancer
Brief Title: ARX788 in HER2-positive Metastatic Breast Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Min Yan, MD, Chief Physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-Breast-09
Record Dates: First submitted 2024-10-23; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: HER2-positive, Metastatic Breast Cancer
Keywords: ARX788; HER2-positive breast cancer; Q6W
MeSH Terms: conditions — Breast Neoplasms | interventions — ARX788

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ARX788 (Experimental)
  Interventions: Drug: ARX788

INTERVENTIONS:
Drug: ARX788 — 2.2 mg/kg IV infusion on Day 1 of each 42-day treatment cycle.

SUMMARY:
A phase 2 study of ARX788 given every 6 weeks in HER2-positive, metastatic breast cancer patients.

DETAILED DESCRIPTION:
A single arm, phase 2 study of ARX788 in HER2-positive, metastatic breast cancer patients. The ARX788 will be administered every 6 weeks (Q6W) intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old (including upper and lower limits), male or female;
* Unresectable locally advanced, recurrent or metastatic BC;
* Has previously received ≤ two lines of chemotherapy (excluding hormone therapy) for recurrent or metastatic BC;
* Tissue samples determined to be HER2 positive (defined as IHC3+ or FISH+);
* Has at least one measurable target lesion as per RECIST1.1 criteria;
* Has recovered from any AE (≤ Grade 1) related to prior surgery and prior cancer treatment;
* Adequate bone marrow, liver, kidney and coagulation function;
* ECOG Performance Status Score of 0-1;
* Voluntarily sign the informed consent, have good compliance and are willing to comply with the follow-up visit.

Exclusion Criteria:

* Has known history to be allergic to any active ingredient or excipient of ARX788;
* With meningeal metastases or disseminated brain metastases or active brain metastases, who need radiation, surgery or drug therapy;
* Has pericardial effusion, pleural effusion or ascites effusion with clinical symptoms, signs or require symptomatic treatment;
* Has interstitial lung disease requiring steroid therapy, a history of drug-induced interstitial lung disease, a history of radiation pneumonitis, or any evidence indicating clinically active interstitial lung disease;
* Has any eye disease that require medical intervention such as keratitis, corneal diseases or active eye infection;
* Has cardiac insufficiency;
* Uncontrolled hypertension;
* Has evidence of severe or uncontrollable systemic diseases;
* Received live vaccines within 4 weeks before the first use of the investigational product or plans to receive live vaccines during the trial;
* Breastfeeding female, or who has childbearing potential with a positive baseline pregnancy test or who is unwilling to use effective contraception during the trial;
* Is unwilling or unable to stop wearing corneal contact lens during the trial;
* Has received any systemic anti-tumor therapy (with the exception of endocrine therapy, with an interval of at least 7 days) within 28 days (or at least 5 half-lives) before the first use of the investigational product;
* Has any mental or cognitive disorder that may restrict his/her understanding and execution of the informed consent form;
* Other conditions that the Investigator considers inappropriate for participation in this trial, such as poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2029-11-20 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | up to 2 years
  ORR is defined as the percentage of participants in the analysis population who have CR or PR per RECIST 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 2 years
  DCR is defined as the percentage of participants in the analysis population who have CR or PR or SD per RECIST 1.1.
Duration of relief (DOR) | From response initiation (when either CR or PR is first determined) to progression or death, whichever occurs first, assessed up to 2 years.
  DOR is defined as the interval from response initiation (when either CR or PR is first determined) to progression or death, whichever occurs first.
Progression-free survival (PFS) | From first dose to first documented disease progression (PD) or death from any cause, whichever occurred first, assessed up to 2 years.
  PFS was defined as the time from first dose to first documented disease progression (PD) or death from any cause, whichever occurred first.
Overall survival (OS) | From the date of first dose of study drug to any-cause death, assessed up to 5 years
  OS was defined as the time from the first dose of study drug to any-cause death.
The number of subjects experiencing adverse event TEAEs | up to 2 years
  Number of participants with TEAEs as assessed by CTCAE v5.0
Pharmacokinetic parameter: Maximum concentration (Cmax) | At the end of Cycle 1 (each cycle is 42 days)
Pharmacokinetic parameter: Time to Cmax (tmax) | At the end of Cycle 1 (each cycle is 42 days)
Pharmacokinetic parameter: Terminal half-life (t1/2) | At the end of Cycle 1 (each cycle is 42 days)
Pharmacokinetic parameter: Area under the concentration-time curve from zero extrapolated to infinity [AUC(0-inf)] | At the end of Cycle 1 (each cycle is 42 days)
Pharmacokinetic parameter: Area under the concentration-time curve from zero to the last quantifiable concentration [AUC(0-last)] | At the end of Cycle 1 (each cycle is 42 days)
Pharmacokinetic parameter: Terminal rate constant (λz) | At the end of Cycle 1 (each cycle is 42 days)
Pharmacokinetic parameter: Systemic clearance (CL) | At the end of Cycle 1 (each cycle is 42 days)
Pharmacokinetic parameter: Volume of distribution (Vz) | At the end of Cycle 1 (each cycle is 42 days)
Pharmacokinetic parameter: Volume of distribution at steady state (Vss) | At the end of Cycle 3 (each cycle is 42 days)
Pharmacokinetic parameter: Trough concentration (Ctrough) | At the end of Cycle 3 (each cycle is 42 days)